CLINICAL TRIAL: NCT06094933
Title: A Randomized Controlled Trial of the Mobile Anger Reduction Intervention for Veterans
Brief Title: Mobile Anger Reduction Intervention
Acronym: MARI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4561-R
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Stress Disorder; Anger
Keywords: posttraumatic stress disorder; anger; hostile interpretation bias; mHealth
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Anger Reduction Intervention (MARI) (Experimental): Participants in this arm will download the MARI application (app) on their own smart phone device and will use the app for a period of 4 weeks.
  Interventions: Behavioral: Mobile Anger Reduction Intervention (MARI)
- Health Education Condition (HED) (Active Comparator): Participants in this arm will download the HED application (app) on their own smart phone device and will use the app for a period of 4 weeks.
  Interventions: Behavioral: Health Education Condition (HED)

INTERVENTIONS:
Behavioral: Mobile Anger Reduction Intervention (MARI) — This is a mobile intervention that uses interpretation bias modification (IBM) techniques to reduce the hostile interpretation bias. Participants will download the MARI app and be instructed to complete at least 5 treatment sessions each week for a period of 4 weeks. Each session takes approximately 10 minutes. The app also includes a Nightly Diary to track symptoms, a calendar to program session reminders, and a My Progress feature to track use and performance.
  Arms: Mobile Anger Reduction Intervention (MARI)
Behavioral: Health Education Condition (HED) — This is a mobile application that delivers videos with psychoeducation about healthy habits and selfcare for general wellness. Participants will download the HED app and be instructed to use it at least 5 times a week for a period of 4 weeks.
  Arms: Health Education Condition (HED)

SUMMARY:
Difficulty controlling anger is the most commonly reported reintegration concern among combat Veterans, especially those with a diagnosis of posttraumatic stress disorder (PTSD). Problematic anger is associated with significant functional impairment. In the current project, the investigators will compare the Mobile Anger Reduction Intervention (MARI) with a health education mobile intervention (HED) among Veterans with PTSD and problematic anger. Participants will be randomized to the MARI or HED condition. The hypothesis is that participants in the MARI condition will experience greater anger reductions and functional improvements relative to the HED condition.

DETAILED DESCRIPTION:
Difficulty controlling anger is the most commonly reported reintegration concern among combat Veterans, especially those with a diagnosis of posttraumatic stress disorder (PTSD). In Veterans, problematic anger is associated with numerous negative psychosocial outcomes, including poor functional outcomes (both social and occupational), family discord, aggression, road rage, and suicide risk. Anger can also impede successful outcomes from PTSD treatment. Given the high prevalence of anger problems among Veterans with PTSD and the associated functional impairments, there is a clear need to develop innovative and effective anger interventions to improve functional outcomes. Use of mobile health (mHealth) technology could provide a low-cost method to increase the reach of anger management treatments to this high-need group of Veterans.

One of the mechanisms associated with problematic anger and aggression is hostile interpretation bias, i.e., a tendency to interpret ambiguous interpersonal situations as hostile. By reducing hostile interpretation bias, the investigators can reduce problematic anger and aggression and improve functional outcomes. A mobile application that uses evidence-based interpretation bias modification techniques to reduce hostile interpretation bias and anger outcomes has been developed and piloted. The goal of this project is to evaluate the efficacy of this mobile application among Veterans with PTSD.

A randomized controlled trial (RCT) will be conducted, in which 150 Veterans with PTSD and problematic anger will be randomized to either the Mobile Anger Reduction Intervention (MARI) or a health education condition (HED). The central hypothesis is that participants in the MARI condition will experience greater anger reductions and functional improvements relative to the HED condition.

The proposed research project will address the following Specific Aims: Aim 1: To evaluate the efficacy of MARI on anger outcomes (e.g., hostile interpretation bias, problematic anger) measured at post-treatment, 3-months, and 6-months post treatment; Aim 2: To evaluate the efficacy of MARI on functional improvements (i.e., psychosocial functioning, quality of life) and self-harm measured at post-treatment, 3-months, and 6-months post treatment; and Exploratory Aim: To explore whether changes in hostile interpretation bias (proposed treatment mechanism) mediate functional improvements.

ELIGIBILITY:
Inclusion Criteria:

* Veterans diagnosed with PTSD, established via chart review and a score of greater than or equal to 33 on the PTSD Checklist for DSM-5 (PCL-5)
* Reporting a score of greater than or equal to 12 on the 5-item Dimensions of Anger Reactions Scale
* Have not had any changes to type or dose of psychiatric medications for 3 months, with no plans to make adjustments in the next 6 months
* Able to read at least 6th grade level material

Exclusion Criteria:

* Currently in a period of active psychosis or mania
* Exhibit current prominent suicidal or homicidal ideation requiring immediate intervention
* Have used the MARI application before as part of another research study
* Receiving (or plan to receive) other anger management psychotherapy or trauma-focused therapy for PTSD (i.e., prolonged exposure, cognitive processing therapy during the course of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
number of participants below the clinical cut off for problematic anger | Post-treatment (approx. one month after baseline assessment)
  Measured with the Dimensions of Anger Reactions-5 scale; scores range from 5-25, with higher scores indicating higher levels of problematic anger; the clinical cut off is 12. The investigators will count the number of participants in each group who have a score lower than 12.
number of participants below the clinical cut off for problematic anger | 6-month follow-up
  Measured with the Dimensions of Anger Reactions-5 scale; scores range from 5-25, with higher scores indicating higher levels of problematic anger; the clinical cut off is 12. The investigators will count the number of participants in each group who have a score lower than 12.
number of participants below the clinical cut off for problematic anger | 3-month follow-up
  Measured with the Dimensions of Anger Reactions-5 scale; scores range from 5-25, with higher scores indicating higher levels of problematic anger; the clinical cut off is 12. The investigators will count the number of participants in each group who have a score lower than 12.
number of participants with decreased hostile interpretation bias scores | from baseline to post-treatment assessments (approx. one month after baseline assessment)
  Measured with the Word Sentence Association Paradigm-Hostility, hostility subscale. Scores range from 1-6, with higher scores indicating higher levels hostile interpretation bias. The investigators will count the number of participants in each group who have a reduction in scores within the time frame.
number of participants with decreased hostile interpretation bias scores | from baseline to 3-month follow-up
  Measured with the Word Sentence Association Paradigm-Hostility, hostility subscale. Scores range from 1-6, with higher scores indicating higher levels hostile interpretation bias. The investigators will count the number of participants in each group who have a reduction in scores within the time frame.
number of participants with decreased hostile interpretation bias scores | from baseline to 6-month follow-up
  Measured with the Word Sentence Association Paradigm-Hostility, hostility subscale. Scores range from 1-6, with higher scores indicating higher levels hostile interpretation bias. The investigators will count the number of participants in each group who have a reduction in scores within the time frame.

SECONDARY OUTCOMES:
number of participants with decreased psychosocial impairment scores | from baseline to post-treatment assessments (approx. one month after baseline assessment)
  Measured with the Brief Inventory of Psychosocial Functioning. Scores range from 0-6, with higher scores indicating higher levels of psychosocial impairment. The investigators will count the number of participants in each group who have a reduction of scores within the time frame.
number of participants with decreased psychosocial impairment scores | from baseline to 3-month follow-up
  Measured with the Brief Inventory of Psychosocial Functioning. Scores range from 0-6, with higher scores indicating higher levels of psychosocial impairment. The investigators will count the number of participants in each group who have a reduction of scores within the time frame.
number of participants with decreased psychosocial impairment scores | from baseline to 6-month follow-up
  Measured with the Brief Inventory of Psychosocial Functioning. Scores range from 0-6, with higher scores indicating higher levels of psychosocial impairment. The investigators will count the number of participants in each group who have a reduction of scores within the time frame.
number of participants with improved quality of life | from baseline to post-treatment assessments (approx. one month after baseline assessment)
  Measured with the Quality of Life Inventory. Scores range from -6-6, with higher scores indicating higher levels of satisfaction with life. The investigators will count the number of participants in each group who have an increase in their score within the time frame.
number of participants with improved quality of life | from baseline to 3-month follow-up
  Measured with the Quality of Life Inventory. Scores range from -6-6, with higher scores indicating higher levels of satisfaction with life. The investigators will count the number of participants in each group who have an increase in their score within the time frame.
number of participants with improved quality of life | from baseline to 6-month follow-up
  Measured with the Quality of Life Inventory. Scores range from -6-6, with higher scores indicating higher levels of satisfaction with life. The investigators will count the number of participants in each group who have an increase in their score within the time frame.
number of participants with reduced suicidal ideation | from baseline to post-treatment assessments (approx. one month after baseline assessment)
  Measured with the Columbia- Suicide Severity Rating Scale, suicidal ideation intensity rating. Scores range from 0-25, with higher scores indicating higher intensity of suicidal ideation. The investigators will count the number of participants in each group who have a decrease in their score within the time frame.
number of participants with reduced suicidal ideation | from baseline to 3-month follow-up
  Measured with the Columbia- Suicide Severity Rating Scale, suicidal ideation intensity rating. Scores range from 0-25, with higher scores indicating higher intensity of suicidal ideation. The investigators will count the number of participants in each group who have a decrease in their score within the time frame.
number of participants with reduced suicidal ideation | from baseline to 6-month follow-up
  Measured with the Columbia- Suicide Severity Rating Scale, suicidal ideation intensity rating. Scores range from 0-25, with higher scores indicating higher intensity of suicidal ideation. The investigators will count the number of participants in each group who have a decrease in their score within the time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten H Dillon, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No